CLINICAL TRIAL: NCT05993481
Title: The Effect of More Frequent Noninvasive Blood Pressure Measurement on the Detection of Intraoperative Hypotension
Brief Title: The Noninvasive Blood Pressure Measurement Effect on the Hypotension
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Collaborators: Bakırkoy Dr. Sadi Konuk Training and Research Hospital (Unknown); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Assoc. Prof. Dr. Yasin Tire, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Study Interval
Record Dates: First submitted 2023-07-27; First posted 2023-08-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hypotension During Surgery
Keywords: Intraoperative Hypotension; Noninvasive Blood pressure measurement; More frequent time interval
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 min. BP (Active Comparator): Clinicians will carry out randomized treatments in coordination with research staff.
  The treatments will be: 1) Ephedrine treatment to maintain intraoperative MAP ≥60 mmHg, delayed resumption of chronic antihypertensive medications as monitoring with 5 min. Blood pressure management. The staff anesthesiologist will administer an ephedrine sulfate injection. An initial dose of 5 to 10 mg given as an intravenous bolus is advised for the treatment of clinically significant hypotension during anesthesia to provide an increase in blood pressure in case of MAP< 60 mmHg. However, the dose of each will be titrated as necessary to reach the target mean arterial pressures.
  Interventions: Diagnostic Test: Blood Pressure Measurement
- 2.5 min. BP (Active Comparator): Clinicians will carry out randomized treatments in coordination with research staff.
  The treatments will be: 2) Ephedrine treatment to maintain intraoperative MAP ≥60 mmHg, delayed resumption of chronic antihypertensive medications as monitoring with 2.5 min. Blood pressure management.
  The staff anesthesiologist will administer an ephedrine sulfate injection. An initial dose of 5 to 10 mg given as an intravenous bolus is advised for the treatment of clinically significant hypotension during anesthesia to provide an increase in blood pressure in case of MAP< 60 mmHg. However, the dose of each will be titrated as necessary to reach the target mean arterial pressures.
  Interventions: Diagnostic Test: Blood Pressure Measurement

INTERVENTIONS:
Diagnostic Test: Blood Pressure Measurement — NIBP measurements will be recorded intraoperatively every 2.5 minutes for the group of 2.5 min. Blood pressure management or every 5 minutes for the other group of 5 min. Blood pressure management after providing randomization before the surgery. A calibrated and time-matched same type of standard anesthetic monitor will be used. The monitor will measure blood pressure and display the mean, systolic and diastolic values.
  All blood pressure measurements will be discontinued before the PACU transfer. Data will be automatically downloaded from the monitor to a computer using a software interface program.

SUMMARY:
Around 300 million surgical operations are performed globally, and of these, 40 to 50 million are performed in the USA. The perioperative period is characterized by hemodynamic instability and, most importantly, hypotension. Intraoperative hypotension is frequent, and the incidence ranges between 5% and 99% during non-cardiac surgery, depending on the definition.

The aim of the study is determined as the relationship between two different time intervals of measurements and time spent hypotensive under harm thresholds in non-cardiac surgery in adults having non-cardiac surgery. Secondarily, it will be determined if more frequent non-invasive blood pressure measurement use decreases postoperative acute kidney injury. Exploratory, it will be evaluated if more frequent non-invasive blood pressure use causes pain or nerve injury in the arms or not.

DETAILED DESCRIPTION:
Around 300 million surgical operations are performed globally, and of these, 40 to 50 million are performed in the USA. The perioperative period is characterized by hemodynamic instability and, most importantly, hypotension. Intraoperative hypotension is frequent, and the incidence ranges between 5% and 99% during non-cardiac surgery, depending on the definition.

Intraoperative hypotension can cause an ischemia-reperfusion injury, manifesting as dysfunction of any vital organ. The kidneys and the heart are the most sensitive organs to be affected. Numerous analyses in diverse non-cardiac surgical populations demonstrate clinically meaningful associations between intraoperative hypotension and myocardial injury, acute kidney injury, serious composite complications, and death. The association between hypotension and various complications seems clear. However, hypotension exposure time provokes acute kidney remains unclear.

Myocardial injury after non-cardiac surgery manifests as an acute increase in the concentration of cardiac biomarkers and occurs in 11.6% of non-cardiac surgeries. Myocardial injury after non-cardiac surgery is also associated with a hypotension period, even with only small biomarker increases. Ischemia-reperfusion injury due to hypotension may substantially contribute to postoperative myocardial injury.

Acute kidney injury (AKI) is defined as creatinine increase and urine output and is well-validated in medical patients. Acute kidney injury reportedly prolongs hospitalization and increases readmissions; it is also associated with increased healthcare costs, sepsis, and mortality. However, most of the data regarding outcomes of acute kidney injury originate from cohorts of hospitalized medical patients, patients admitted to critical care units, or trauma victims. Postoperative kidney injury can increase after surgery because of dehydration or surgical muscle injury. Furthermore, a recent study found a strong relationship between intraoperative hypotension exposure and non-cardiac surgery-related acute kidney injury in patients <60 years of age. However, another study found no independent association between varying ages and postoperative acute kidney injury without evaluating intraoperative hypotension exposure.

The definition of intraoperative hypotension is that a mean arterial pressure (MAP) of 65 mm Hg is accepted as a threshold predicting myocardial injury, which is a leading cause of 30-day postoperative mortality. Additionally, the risk of end-organ dysfunction increases with the length of low arterial blood pressure. According to Walsh et al., as little as 1 minute of exposure to MAP <55 mm Hg is associated with myocardial injury, any cardiac complication, and kidney injury after non-cardiac surgery.

The American Society of Anesthesiologists (ASA) "Standards for Basic Anesthetic Monitoring" require measurement and evaluation of arterial blood pressure (BP) at least every five minutes except "under extenuating circumstances," but acknowledge that "brief interruptions of continual monitoring may be unavoidable." The standards apply to all patients undergoing anesthetics (general, regional, or monitored anesthesia care). Intraoperative blood pressure can be measured oscillometrically, usually at 5 minutes intervals, or continuously with an arterial catheter. However, when patients are hemodynamically unstable, the non-invasive blood pressure measurement interval of 5 minutes may be insufficient to assess rapidly changing hemodynamics accurately. Subsequently, the provider sometimes inadvertently fails to re-engage the cyclic measurement of cuff blood pressure. This leads to extended periods when hypotension is not measured, thus potentially compromising patient safety.

Arterial catheters are generally used to monitor hemodynamic fluctuations for certain complex operations and patients with significant comorbidities. Recent studies even suggest that only a few minutes of hypotension in the acute care setting increases the incidence of complications. These observations strongly suggest that continuous blood pressure monitoring is critical in the acute care setting to identify periods of hypertension and/or hypotension as early as possible. Today, the gold standard for blood pressure monitoring is the invasive arterial line, a catheter inserted into an artery, which enables continuous blood pressure monitoring.

On the other hand, it is impossible to place the arterial catheter on all patients because of invasiveness and complications. One extensive study on the topic, in a systematic review, assessed the complications associated with an arterial catheter in >25 000 cases. In this study, temporary artery occlusion was the most frequent complication ranging from 1.5 to 35% (average: 19.7%). Hematomas were the second most common complication, with an incidence of 14.4%. Serious complications such as permanent occlusion, pseudoaneurysm, and sepsis occurred in 0.09%, 0.09%, and 0.13% of cases, respectively.

Therefore, the aim of the study will be determined as the relationship between two different time intervals of measurements and time spend hypotensive under harm thresholds in non-cardiac surgery in adults having non-cardiac surgery. Secondarily, it will be determined if more frequent non-invasive blood pressure measurement use decreases postoperative acute kidney injury. Exploratory, it will be evaluated if more frequent non-invasive blood pressure use causes pain or nerve injury in the arms or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. ASA Physical Status 1 and 3;
3. Non-cardiac surgery with expected surgery duration ≥ 2 hours;
4. Supine position during the surgery;
5. Regional or general anesthesia;
6. Planned hospital stay time of at least 24 hours.

Exclusion Criteria:

1. Patients who confirm to be pregnant and/or nursing mothers;
2. Patients with an intra-aortic balloon pump (IABP) or ventricular assist device(s);
3. Has a condition that precludes routine or tight blood pressure management;
4. Mean arterial blood pressure differences between right and left arm ≥ 5 mmHg;
5. Patient who has physically disabled their arms:

5. Emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The time-average spend hypotensive (under MAP thresholds of 65 mmHg) for at least 1 minute | Every 2.5 minute in the surgery upto end of the surgery.
  For the primary outcome, clinically important difference will be the time-average spend hypotensive (under MAP thresholds of 65 mmHg) for at least 1 minute since it has been shown clinically important in previous studies . We will assess this primary outcome in adults having non-cardiac surgery, a 2.5-minute interval of intraoperative blood measurement group compared to the standard 5-minute interval group.

SECONDARY OUTCOMES:
the time-average spend hypotensive (under MAP thresholds of <60, <50, and <40 mmHg [mmHg]) for at least 1 minute. | Every 2.5 minute in the surgery upto end of the surgery.
  For the secondary outcomes, clinically important difference will be the time-average spend hypotensive (under MAP thresholds of <60, <50, and <40 mmHg [mmHg]) for at least 1 minute, and absolute [n] and relative [%] number of patients with any MAP measurement <65, <60, <50, and <40mmHg, absolute [n] and relative [%] number of patients with at least one 1-minute episode of a MAP <65, <60, <50, and <40 mmHg, time-weighted average MAP >100, >110, >120, >140mmHg [mmHg], time-weighted cumulative amount of ephedrine indexed to body weight [µg kg-1 min-1], cumulative amount of administered fluids indexed to surgical duration [mL min-1]

OTHER OUTCOMES:
Postoperative complications after surgery including acute myocardial infarction, acute kidney injury, non-fatal cardiac arrest, peripheral nerve injuries, arm pain and death and delrium status. | Postoperative time until 24th hours.
  The exploratory outcomes will be Postoperative complications after surgery including acute myocardial infarction, acute kidney injury, non-fatal cardiac arrest, peripheral nerve injuries, arm pain and death, a 2.5-minute interval group of intraoperative blood measurement compared to the standard 5-minute interval group, 2 hours after surgery in the post-anesthesia recovery unit and after 24 hours. And delirium status in person for 24th hours and through the 48th hours (after discharge by phone calling) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Tire, Assoc. Prof., Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Meram, Turkey (Türkiye)